CLINICAL TRIAL: NCT03199950
Title: Delirium: Is Prophylactic Drug Therapy Useful in High Risk Patients as Defined by the Delirium Risk Prediction Model?
Brief Title: PROfylactic Haloperidol in Patients Defined as High Risk for DElirium With Delirium Risk mOdel
Acronym: PRODEO
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zuyderland Medisch Centrum (Other)
Responsible Party: Principal Investigator, Hugo Van der Kuy, Principle Investigator, Zuyderland Medisch Centrum
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 17-T-31; 2017-001260-37 (EudraCT Number)
Record Dates: First submitted 2017-06-23; First posted 2017-06-27 (Actual); Last update posted 2017-06-27 (Actual); Status verified 2017-06

CONDITIONS: Delirium
Keywords: Delirium; Haloperidol; Prophylactic; High-risk
MeSH Terms: conditions — Delirium | interventions — Haloperidol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prophylactic Haloperidol arm (Experimental): Patients will receive oral haloperidol 2dd1mg (08.00am & 10.00pm)
  Interventions: Drug: Haloperidol
- No treatment (Placebo Comparator): Patients will receive oral placebo 2dd (08.00am & 10.00pm)
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Haloperidol — Haloperidol 2dd1mg (08.00am - 10.00pm)
  Other Names: Haldol; RVG 55776
  Arms: Prophylactic Haloperidol arm
Drug: Placebo Oral Tablet — Placebo oral 2dd (08.00am - 10.00pm)
  Arms: No treatment

SUMMARY:
The hospital pharmacy at the Zuyderland Medical Centre developed the DElirium MOdel (DEMO) to predict which patients are at risk of developing a delirium in patients aged 60 or older. With this delirium risk prediction model we aim to predict more accurately which patients are at high risk of developing a delirium and want to investigate if these patients can benefit from prophylactic haloperidol.

DETAILED DESCRIPTION:
Intro: Delirium is a common postoperative complication within geriatric patients. It is described delirium as a very stressful experience for the patient which can lead to prolonged hospital stay, higher cost, additional morbidity and increased mortality.

In 2013 the hospital pharmacy at the Zuyderland Medical Center developed the delirium risk prediction model to determine the chance of development of a delirium in patients aged 60 or older. Electronically available data such as age, polypharmacy, use of anti-dementia drugs, anti-depressants, anti-parkinsonian drugs, anti-diabetics, analgesics and/or sleeping medication were used in the study. The delirium risk prediction model was validated prospectively after retrospective development. The model will be used in this study to predict the risk of developing delirium postoperatively.

We expect prophylactic haloperidol to be effective in patients with a high risk of developing a delirium according to the delirium risk prediction model.

Aim: The PRODEO-study aims to reduce the incidence of postoperative delirium by administering prophylactic haloperidol to patients with a high risk of developing delirium according to the delirium risk prediction model.

Methods: The study is a randomized and double blind single center study with two parallel groups. Subjects ≥60 years with increased risk of postoperative delirium according to the delirium risk prediction model undergoing elective chirurgical or elective orthopedic surgery are eligible. Subjects will be excluded if they already use anti-psychotic drugs, are not able to take oral medication or when there are contra-indications. Haloperidol (1mg) or placebo will be administered at set times postoperatively. Subjects receive haloperidol 2dd1mg or a placebo 2dd during a maximum of five days during admission. On day 3 blood samples will be obtained in order to determine the true concentration levels of haloperidol. The primary endpoint is delirium incidence within 5 days after surgery. Secondary endpoints are costs of treatment, number of admission days, adverse events, true concentration levels of haloperidol and duration and severity of delirium.

Results: The study will start in June 2017 with an inclusion rate of 20 patients per week. An incidence reduction of 30% in the intervention group is expected. To reach sufficient statistical power a study population of 1366 subjects is needed. Duration of the inclusion period is expected to be 18 months.

ELIGIBILITY:
Inclusion criteria

* Age >60 years
* Planned elective surgery
* General surgery or orthopaedic surgery
* At least one night postsurgical admission
* High-risk developing delirium according to the DEMO-model
* Absence of delirium pre-operatively

Exclusion criteria

* Less than 1-day postoperative admission in hospital
* Hypersensitivity to butyrophenone derivates
* Use of antipsychotics
* Not being able to take oral medication
* Presence of contraindications (lesions of basal ganglia, clinical significant heart disease (eg. recent acute myocardial infarction, non-compensated heart failure, arrythmias treated with drugs out of the NYHA(New York Heart Association)-class Ia and II anti-arrythmics), known prolongation of the QT interval, history of ventricular arrythmia and torsades de pointes, uncorrected hypokalemia.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1366 (Estimated)
Dates: Start 2017-06-23 (Actual); Primary Completion 2018-11-23 (Estimated); Study Completion 2018-11-23 (Estimated)

PRIMARY OUTCOMES:
Occurence of delirium | Delirium within 5 days postoperative
  Will prophylactic haloperidol in high risk patients as established with DEMO reduce the incidence of delirium?

SECONDARY OUTCOMES:
Costs of treatment | up to 2 years
  Total costs of hospital stay
Days admitted to hospital | an average of two weeks
  Total amount of days admitted to the hospital
Adverse events of intervention medication | an average of two weeks
  Adverse events during admission in the hospital
Circulating concentration of Haloperidol | up to 2 years
  Blood sample collection at day, trough concentration haloperidol in blood sample
Duration of delirium | an average of two weeks
  Days DOS (Delirium observation scale) positive after surgery,
Severity of delirium | an average of two weeks
  DOS scores during admission

CONTACTS AND LOCATIONS:
Overall Officials: Hugo van der Kuy, Principal Investigator — Zuyderland MC
Locations (1):
- Zuyderland Medisch Centrum, Sittard, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Inouye SK, Studenski S, Tinetti ME, Kuchel GA. Geriatric syndromes: clinical, research, and policy implications of a core geriatric concept. J Am Geriatr Soc. 2007 May;55(5):780-91. doi: 10.1111/j.1532-5415.2007.01156.x. PMID 17493201
- [Background] Demeure MJ, Fain MJ. The elderly surgical patient and postoperative delirium. J Am Coll Surg. 2006 Nov;203(5):752-7. doi: 10.1016/j.jamcollsurg.2006.07.032. Epub 2006 Sep 26. No abstract available. PMID 17084339
- [Background] Salluh JI, Wang H, Schneider EB, Nagaraja N, Yenokyan G, Damluji A, Serafim RB, Stevens RD. Outcome of delirium in critically ill patients: systematic review and meta-analysis. BMJ. 2015 Jun 3;350:h2538. doi: 10.1136/bmj.h2538. PMID 26041151
- [Background] Leslie DL, Marcantonio ER, Zhang Y, Leo-Summers L, Inouye SK. One-year health care costs associated with delirium in the elderly population. Arch Intern Med. 2008 Jan 14;168(1):27-32. doi: 10.1001/archinternmed.2007.4. PMID 18195192
- [Background] Fukata S, Kawabata Y, Fujisiro K, Katagawa Y, Kuroiwa K, Akiyama H, Terabe Y, Ando M, Kawamura T, Hattori H. Haloperidol prophylaxis does not prevent postoperative delirium in elderly patients: a randomized, open-label prospective trial. Surg Today. 2014 Dec;44(12):2305-13. doi: 10.1007/s00595-014-0859-7. Epub 2014 Feb 16. PMID 24532143
- [Background] Wang W, Li HL, Wang DX, Zhu X, Li SL, Yao GQ, Chen KS, Gu XE, Zhu SN. Haloperidol prophylaxis decreases delirium incidence in elderly patients after noncardiac surgery: a randomized controlled trial*. Crit Care Med. 2012 Mar;40(3):731-9. doi: 10.1097/CCM.0b013e3182376e4f. PMID 22067628
- [Background] de Wit HA, Winkens B, Mestres Gonzalvo C, Hurkens KP, Mulder WJ, Janknegt R, Verhey FR, van der Kuy PH, Schols JM. The development of an automated ward independent delirium risk prediction model. Int J Clin Pharm. 2016 Aug;38(4):915-23. doi: 10.1007/s11096-016-0312-7. Epub 2016 May 13. PMID 27177868